CLINICAL TRIAL: NCT03855111
Title: Symptom Management Efficacy Study to Reduce Distal Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S18-00257; NIH-1R01NR017917-01 (Other Grant/Funding Number: National Institutes of Health)
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain; HIV Neuropathy; HIV/AIDS; Pain
Keywords: Neuropathic pain; HIV Neuropathy; HIV/AIDS; Symptom Management; Acupuncture; Pain; Pain Syndrome
MeSH Terms: conditions — Neuralgia; Acquired Immunodeficiency Syndrome; Pain; Somatoform Disorders | interventions — Moxibustion

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, placebo-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard (fixed) protocol Acu/Moxa - Active (Experimental): Standard (Fixed) Acupuncture / Moxibustion Active Protocol
  Subjects receive active standard Acu/Moxa protocol aimed at reducing neuropathic pain/discomfort.
  Interventions: Other: Standard Acupuncture / Moxibustion
- Individualized (tailored) protocol Acu/Moxa - Active (Experimental): Individualized (Tailored) Active Acupuncture / Moxibustion Protocol
  Subjects receive active individualized Acu/Moxa protocol based on traditional Chinese medicine assessment aimed reducing neuropathic pain/discomfort.
  Interventions: Other: Individualized (Tailored) Active Acupuncture / Moxibustion
- Sham Acu/Placebo Moxa (Control) (No Intervention): Sham Acu/Placebo Moxa (Control)
  Note. All subjects randomized to the Control will be offered 12 active protocol acupuncture/ moxibustion treatments, at no cost, at the end of their study participation.
- WaitList (Control) (No Intervention): WaitList (Control) No treatment. Subjects receive all aspects of study participation with the exception of exposure to Acupuncture / Moxibustion.
  Note. All subjects randomized to the Control will then be offered 12 active protocol acupuncture/ moxibustion treatments, at no cost, at the end of their study participation.

INTERVENTIONS:
Other: Standard Acupuncture / Moxibustion — Standard (Fixed) Active Acupuncture / Moxibustion protocol aimed at reducing lower limb neuropathic pain/discomfort.
  Other Names: Standard Acupuncture /Moxibustion
  Arms: Standard (fixed) protocol Acu/Moxa - Active
Other: Individualized (Tailored) Active Acupuncture / Moxibustion — Individualized (tailored) protocol Acu/Moxa - Active. Acu/Moxa prescription based on TCM assessment. Protocol aimed at reducing lower limb neuropathic pain/discomfort.
  Other Names: Individualized Active Acupuncture / Moxibustion
  Arms: Individualized (tailored) protocol Acu/Moxa - Active

SUMMARY:
Distal sensory peripheral neuropathy (DSP) is a chronic, debilitating painful condition affecting quality of life in persons living with HIV. Treatments prescribed to manage DSP pain, such as nonnarcotic and narcotic analgesics, antidepressants and anticonvulsants, are largely ineffective. In HIV there are no FDA-approved drugs for this indication. This study assesses in a randomized controlled clinical trial, the efficacy of novel non-pharmacologic pain management approaches to reduce HIV-related DSP pain and improve quality of life.

DETAILED DESCRIPTION:
Distal sensory peripheral neuropathy (DSP) is a chronic, debilitating painful condition affecting quality of life in 20%-50% of persons living with HIV. Treatments prescribed to manage DSP pain, such as nonnarcotic and narcotic analgesics, antidepressants and anticonvulsants, are largely ineffective. Effective management of DSP pain is an unmet therapeutic need for this population. This study is a randomized, blinded, placebo-controlled clinical trial of the efficacy of Acupuncture/Moxibustion (Acu/Moxa) for HIV DSP pain/discomfort.

Subjects with HIV-related lower limb DSP pain are randomized to one of four Conditions: 1) Standard (fixed) protocol Acu/Moxa, 2) Individualized (tailored) protocol Acu/Moxa, 3) Sham Acu/Placebo Moxa (control), or 4) WaitList (control). Subjects attend six weeks of twice weekly treatment sessions and 3 non-treatment follow-up sessions at weeks 9, 11, and 15. All subjects are assessed by a blinded diagnostic acupuncturist (DA) and those assigned to Conditions 1, 2 and 3 receive treatments by an unblinded treating acupuncturist (TA). Specific Aims are: #1 determine group differences in weekly average pain (Gracely Pain Scale) at the end of treatment (Tx) and end of follow-up (F/U); SA#2 determine group differences in improvement in specific sensory symptoms (Subjective Peripheral Neuropathy Screen and neurological sensory testing (NST)) and patient-rated effectiveness (Clinical Global Improvement, NIH PROMIS Pain Intensity and Health-Related Quality of Life (MOS-HIV)) at Tx and F/U; SA#3 determine group differences in safety profiles; and SA#4, explore how baseline measures, TCM diagnoses, NST and pain medication use predict response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older, HIV+ or AIDS diagnosed, with a history of DSP of the lower extremities for the past three months or greater.
* Primary care provider (PCP) verification of HIV status, diagnosis of DSP, & subject clinical suitability for the study.
* Evidence of lower limb neuropathy (bilateral ankle reflexes absent or depressed relative to the knee, decreased sensation to vibration, pin prick and temperature with distal sensory loss grading to normal in the proximal limb)
* GPS rated pain severity of "moderate" or above, documented in 1-week prospective self-report symptom diary (SD).
* Any antiretroviral Rx must have 3 months of stable regimen (same drugs, dose & frequency) prior to enrollment.
* Any pain medications must have 3 months of stable regimen prior to enrollment.
* Those on a stable pharmacologic regimen are expected to remain on the regimen for the duration of the study.
* Must understand and agree to complete daily symptom diaries for the duration of the study.
* Successfully complete a mini-mental status exam (obtaining a score of 24 or above).

Exclusion Criteria:

* Any acute condition requiring medical care (eg. opportunistic infection).
* Conditions that may mimic HIV DSP symptoms: i.e. diabetes(3), coagulopathies, B12 deficiency, etc.
* Use any topically applied medications to the lower extremities.
* Alcohol and/or substance dependence.
* Use of injectable corticosteroids or any medications known to be neurotoxic within 3 months prior to enrollment.
* Pregnant women or unwilling to use an acceptable form of birth control.
* Receiving acupuncture within 6 months prior to enrollment.
* Any history of receiving moxibustion.
* Currently receiving any other complementary therapies such as herbs, massage, reiki etc.
* Relocation or plans that interfere with attending all of the planned study sessions and/or recording SD information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Gracely Pain Scale (GPS) | Change from baseline rating of pain/discomfort (Gracely Pain Scale) after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine sustainability).
  The GPS is a Likert magnitude-estimation log-scale of sensory pain. Subjects rate their DSP pain by selecting one of 13 words to describe their average and worst DSP pain.
  "Nothing"=0 to "Extremely intense"=12

SECONDARY OUTCOMES:
Subjective Peripheral Neuropathy Screen (SPNS) | Change from baseline rating of neuropathy symptoms after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine change and sustainability)
  Describes neuropathy symptoms eg. aching/burning, "pins and needles", numbness, location (hands/arms, feet/legs), and severity of symptoms from "minimal" to "extreme".
NIH PROMIS Pain Scale | Change from baseline rating of pain intensity after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine change and sustainability)
  NIH Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity short form is used to assess "how much a person hurts". Subjects in the last 7 days, the worst pain intensity, the average pain intensity. Subjects rate their pain intensity from none (=1) to very severe (=5).
Medical Outcome Survey - HIV (MOS-HIV) | Change from baseline rating of general health after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine change and sustainability)
  General health-related quality of life questions in HIV that assesses ten dimensions of health (overall health, pain, physical functioning, role and social functioning, mental health, energy/fatigue, cognitive function, health distress
Clinical Global Severity Improvement Scale (CGIs) | Change from baseline rating of pain intensity after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine change and sustainability)
  The severity of illness scale measures global severity of symptoms [in the context of peripheral neuropathy]. The patient rates discomfort from peripheral neuropathy on a scale of 0= No discomfort to 6= Very severe discomfort. The global improvement component measures the level of change from initial severity: 0= No improvement at all to 6= Great improvement
Neurological Sensory Testing (NST) | Change from baseline neurological physical assessment after 6 wks of twice-wkly treatment sessions (the end of the treatment phase) and at weeks 9, 11 and 15 (the follow-up phase - determine change and sustainability)
  Neurological assessments with Neuro Sensory Testing (NST) include: muscle strength and reflexes and sensory testing for lower limb vibration, pain and thermal sensation. Standard neurological assessment: muscle strength 0-5; reflexes 0-5; pain- intact, reduced, absent, hyperalgesia; vibration - intact, impaired; thermal - intact, reduced absent. The neuro/NST also serves to monitor for clinical safety and findings.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, Division of Special Studies in Symptom Management, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Congruent with NIH policy, the PI will make any unique resources e.g. the protocol and materials developed for this research study be available for research purposes to qualified individuals within the scientific community through publication and presentations. In addition, research information will be made available upon request to Dr. Joyce K. Anastasi.
Supporting Information: Study Protocol, CSR
Time Frame: After the outcome paper has been published
Access Criteria: Contact Principal Investigator